CLINICAL TRIAL: NCT05702554
Title: Recruitment-to-inflation Ratio to Set Positive End-expiratory Pressure for Laparoscopic/Robotic Surgery: a Multicenter Study
Acronym: PEEP_LAP1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera di Perugia (Other)
Responsible Party: Principal Investigator, Prof Gianmaria Cammarota, Prof Gianmaria Cammarota, Azienda Ospedaliera di Perugia
Other Study IDs: PEEP_LAP1
Record Dates: First submitted 2023-01-19; First posted 2023-01-27 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Respiratory System Mechanics; Pneumoperitoneum
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present investigation is focused to assess the effects of positive end-expiratory pressure (PEEP) on respiratory system compliance in obese patients invasive mechanical ventilation for laparoscopic or robotic surgery with pneumoperitoneum

DETAILED DESCRIPTION:
Adult obese (body mass index ≥ 30 kg/m2) patients undergoing invasive mechanical ventilation for laparoscopic or robotic surgery with pneumoperitoneum will be enrolled, upon the acquisition of informed consent.

Will be excluded all the patients with the following conditions: American society of anesthesiologists (ASA) score ≥ 4; severe cardiopathy, intracranial hypertension, tracheostomy, previous cardio-thoracic surgery, pulmonary hypertension, broncho-pleural fistula, pulmonary emphysema, pneumothorax, chronic respiratory failure, chronic obstructive pulmonary disease, pregnancy.

Thereafter, general anesthesia will be induced, according to current clinical practice and mechanical ventilation will be commenced according to current recommendations.

Following the application of definitive pneumoeritoneum and body position, the recruitment/inflation procedure will be carried out to identify PEEP. PEEP-induced recruitment will be computed with high PEEP set at 15 cmh2o (or higher) and low PEEP set at 5 cmh2o. In case of an airway opening pressure > 5 cmh2o, the airway opening pressure (AOP) will be set as low PEEP and the high PEEP will be set at the value corresponding to AOP+ 10 cmh20. During the procedure, tidal volume will be maintained between 6-8 ml/kg of predicted body weight. On the basis of the recruitment-to-inflation ratio (R/I), PEEP will be set as follows: low PEEP, in presence of R/I < 0,5; high PEEP with R/I ≥ 1.5; PEEP set within low and high PEEP range on clinical decision, if R/I ≥ 0.5 and <1.5.

After 20 min from the onset of mechanical ventilation and 1 hour from PEEP application following pneumoperitoneum and definitive body position, mechanics of the respiratory system for compliance and driving pressure will be assessed.

As an optional evaluation, a lung ultrasound examination will be performed before general anesthesia induction and 1 hour after extubation, before discharging the patient from recovery room.

During anesthesia vital signs will be continuously monitored. On the clinically judgement, arterial blood gases will be carried out across the study stages.

ELIGIBILITY:
Inclusion Criteria:

* Adult obese (body mass index ≥ 30 kg/m2) patients undergoing invasive mechanical ventilation for laparoscopic or robotic surgery with pneumoperitoneum will be enrolled, upon the acquisition of informed consent.

Exclusion Criteria:

* Will be excluded all the patients with the following conditions: american society of anesthesiologists (ASA) score ≥ 4; severe cardiopathy, intracranial hypertension, tracheosthomy, previous cardio-thoracic surgery, pulmonary hypertrension, broncho-pleural fistula, pulmonary emphysema, pnumothorax, chronic respiratory failure, chronic obstructive pulmonary disease, pregnancy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult obese (body mass index ≥ 30 kg/m2) patients undergoing invasive mechanical ventilation for laparoscopic or robotic surgery with pneumoperitoneum
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-08-05 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative respiratory system mechanics | 1 hour following PEEP application
  respiratory system compliance defined as volume variation to pressure variation ratio

SECONDARY OUTCOMES:
respiratory pulmonary complications incidence | up to 7 days after surgery
  the number of pulmonary complications (hypoxaemia with oxygen saturation less than or equal to 92% requiring suplemental oxygen administration, atelectasis, pneumothorax, pneumonia, acute respiratory distress syndrome, reintubation

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Università degli Studi di Perugia, Perugia, Umbria, Italy
  - Università degli Studi di Perugia, Perugia